CLINICAL TRIAL: NCT07081581
Title: Comparison of the Postoperative Analgesic Efficacy of Serratus Plane Block With Different Adjuvant Agents in Breast Cancer Surgery
Brief Title: Analgesic Effect of Serratus Plane Block With Adjuvant Agents in Breast Cancer Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Dilek Yamac, specialist doctor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBU-ANESTEZİ-DMY-03
Record Dates: First submitted 2025-06-08; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Post Operative Pain
Keywords: pain management; serratus anterior plane block; Breast cancer surgery
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Agnosia | interventions — Bupivacaine; Control Groups; Magnesium Sulfate; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: After induction of general anaesthesia, serratus anterior plane block was performed in all patients. Group B received bupivacaine (control group), Group D received bupivacaine + dexmedetomidine, Group M received bupivacaine + magnesium sulphate.
Who Masked: Participant, Care Provider
Masking Description: Drugs administered in regional blocks were prepared according to group randomisation by an anaesthetist not involved in patient management or data collection. Patients were divided into three groups using a sealed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group B (Experimental): Group B (Blockade with Bupivacaine): 30 mL bupivacaine (0.25%)
  Interventions: Drug: Bupivacain
- Group M (Experimental): Group M (Bupivacaine+Magnesium Blockade): 30 mL bupivacaine (0.25%) + 500 mg magnesium sulphate
  Interventions: Drug: Bupivacaine and Magnesium sulfate
- Group D (Experimental): Group D (bupivacaine + dexmedetomidine ile Blokaj): 30 mL bupivacaine (% 0.25) + 1 μg/kg dexmedetomidine.
  Interventions: Drug: Bupivacaine and Dexmedetomidine ile Blokaj

INTERVENTIONS:
Drug: Bupivacain — In Group B( control group), bupivacaine was given as additional medication in the serratus block application.
  Other Names: Control group
  Arms: Group B
Drug: Bupivacaine and Magnesium sulfate — In Group M, bupivacaine and magnesium were given as additional medication in the serratus block application.
  Other Names: Local anesthetic with added adjuvant agent(1)
  Arms: Group M
Drug: Bupivacaine and Dexmedetomidine ile Blokaj — In Group D, bupivacaine and dexmedetomidine were given as additional medication in the serratus block application.
  Other Names: Local anesthetic with added adjuvant agent(2)
  Arms: Group D

SUMMARY:
Pain after breast surgery has been described as moderate to severe in intensity and, if inadequately treated, increases postoperative morbidity, hospital cost, and the incidence of persistent postoperative pain. Serratus anterior plane block is an interfascial injection technique for analgesia of the chest wall. The aim of this study was to investigate the effect of magnesium and dexmedetomidine as adjuvant agents on postoperative analgesia in serratus anterior plane block in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
In this prospective, double-blind, randomised controlled study, a total of 75 patients aged 30-70 years, who were planned for elective modified radical mastectomy after ethics committee approval, were included. Patients were randomly divided into three groups. After induction of general anaesthesia, serratus anterior plane block was applied to all patients. Group B received bupivacaine 30 ml (0.25%), Group D received bupivacaine 30 ml (0.25%) + dexmedetomidine 1μg/kg, Group M received bupivacaine 30 ml (0.25%) + 500 mg magnesium sulphate. Haemodynamic parameters, numerical rating scale (NRS) scores, number of tramadol use with patient-controlled analgesia device, additional analgesic drug consumption and side effects were recorded at 2, 6, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria: - 30-70 years old, ASA I-II-III patient group,

* Not hypersensitive to the drugs to be used in the study or to the substances contained in them,
* No infection or anatomical deformation at the site of intervention,
* No antithrombotic treatment and normal coagulation parameters,
* Patients who have the consent of themselves or one of their legal guardians.

Exclusion Criteria:

* Less than 30 years of age, older than 70 years of age or ASA (American Society of Anaesthesiologists) Classification IV,
* Receiving antithrombotic therapy with abnormal coagulation parameters,
* Infection or anatomical abnormality at the blockage site,

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic efficacy | until the 24th hour postoperatively
  Hemodynamic parameters (heart rate, noninvasive mean arterial blood pressure, peripheral oxygen saturation), numerical rating scale (NRS) scores, number of tramadol uses with patient-controlled analgesia device, and additional analgesic drug consumption were recorded at 2, 6, 12, and 24 hours after surgery. The Numerical Rating Scale (NRS) is a subjective scale in which patients rate their pain intensity by selecting a number between 0 and 10. 0 means "no pain," while 10 means "worst pain imaginable." Patients typically rate their pain over the past 24 hours. It can be used in both verbal and written formats.

SECONDARY OUTCOMES:
Complications due to adjuvant agents | until the 24th hour postoperatively
  Complications due to adjuvant agents used in serratus plan blockade

CONTACTS AND LOCATIONS:
Overall Officials: Dilek MD Metin Yamac, Principal Investigator — Sultan Abdülhamid Han education and research hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No